CLINICAL TRIAL: NCT06170749
Title: Prediction Model for Anemia After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other); Jining First People's Hospital (Other); The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yuntao Nie, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: CJBariatric003
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Anemia; Bariatric Surgery
Keywords: Anemia; Bariatric surgery; Prediction model
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop and validate a prediction model for estimating the short and long-term risk of anemia after bariatric surgery.

DETAILED DESCRIPTION:
This study aims to develop and validate a prediction model for estimating the probability of anemia for patients with obesity one, three, and five years after sleeve gastrectomy and Roux-en-Y gastric bypass, using preoperative clinical and laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* aged between 16-70 years;
* body mass index (BMI) ≥ 27.5 kg/m2;
* complete preoperative and follow-up data.

Exclusion Criteria:

* vegetarian;
* other bariatric procedures;
* renal failure at baseline;
* postoperative bleeding (it was defined as a drop in hemoglobin levels > 3 g/dL or a confirmed blood loss requiring treatment after surgery);
* incomplete preoperative and follow-up data.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study aims to include patients with obesity who will undergo bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
AUCs of the prediction model at 1, 3, 5 years | 5 years
  This metric shows the discrimination ability of the prediction model.

SECONDARY OUTCOMES:
Brier score | 5 years
  This metric shows the calibration of the model. The Brier score (on a scale ranging from 0 to 1), which calculates the difference between the estimated and observed risk for malignancy with values closer to 0 indicating better calibration, was used to evaluate model calibration.

OTHER OUTCOMES:
AUCs of the prediction model in different subgroups | 5 years
  AUCs of the prediction model in different subgroups, including age (≤ 40 years/>40 years), sex, BMI (≤37.5kg/m2/>37.5kg/m2), smoking history, alcohol consumption, hypertension, and T2DM history.

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Nie, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Yuntao Nie, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to the medical privacy implications of the study data, the principal investigator needs to be contacted for access.